CLINICAL TRIAL: NCT00059527
Title: Youth Environments Promoting Nutrition and Activity
Brief Title: Healthy Youth Places: A Program to Promote Nutrition and Physical Activity in Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5R01HD37367-3; 5R01HD037367 (NIH)
Record Dates: First submitted 2003-04-28; First posted 2003-04-29 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2005-08

CONDITIONS: Health Behavior
Keywords: Physical Activity; Nutrition; Self Efficacy; Middle School; Intervention
MeSH Terms: conditions — Health Behavior; Motor Activity

INTERVENTIONS:
Behavioral: Healthy Youth Places: a behavior change model

SUMMARY:
To reduce the risk for chronic disease, adolescents should eat at least five servings of fruit and vegetables and be physically active daily. This study will implement and evaluate a school-based program to encourage adolescents to achieve and maintain a healthy diet and exercise regimen.

DETAILED DESCRIPTION:
The Healthy Youth Places project will test if an intervention strategy that implements school environmental change, with both adult leader and youth participation, will influence and maintain adolescent fruit and vegetable consumption and physical activity.

The study will assess the effects of school environment and curriculum interventions promoting fruit and vegetable (F&V) consumption, physical activity (PA), and their environmental determinants. The project will involve goal-setting and efficacy-building interventions designed to develop the skills and group efficacy of both adult school personnel and students. The adult-based interventions are designed to change the school environments through a school coalition assisted by a local coordinator. The youth interventions involve the participation of students in the processes of building the local health behavior environments and target both school lunch and after-school activity environments.

The project encourages adult and youth participation in the process of planning and implementing environmental change in targeted adolescent physical and social environments (school lunch place, after-school program place). Environmental change is defined as implemented practices, programs, and policies that promote critical elements (connection, autonomy, skill-building, healthy fruit and vegetable and physical activity norms). These critical elements are social environmental processes of behavior change.

Sixteen schools will be randomly assigned to either the experimental or the control (no treatment) condition. The health behavior of adolescents will be assessed during the sixth, seventh, eighth, and ninth grades. Measurement of F&V and PA behaviors are the primary outcomes and will be assessed by self-report and verified by objective measures of school lunch purchases and physical activity monitoring. The impact of the program on personal, environmental, and behavioral determinants of F&V and PA will also be measured.

ELIGIBILITY:
Inclusion Criteria

* Student attending sixth through eighth grades
* Participating middle school

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000
Dates: Start 1999-03; Study Completion 2003-05

PRIMARY OUTCOMES:
Moderate and Vigorous Physical Activity
Vigorous Physical Activity
Fruit and Vegetable Consumption

SECONDARY OUTCOMES:
Self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: David A Dzewaltowski, Ph.D., Principal Investigator — Community Health Institute, Kansas State University

REFERENCES:
- [Background] Dzewaltowski DA, Estabrooks PA, Johnston JA. Healthy youth places promoting nutrition and physical activity. Health Educ Res. 2002 Oct;17(5):541-51. doi: 10.1093/her/17.5.541. PMID 12408199
- See also: Click here for more information about the intervention framework — http://www.healthyplaces.org
- See also: Click here for more information about the evaluation framework — http://www.re-aim.org